CLINICAL TRIAL: NCT00578058
Title: Randomized Trial Of Tinnitus Retraining Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Richard S. Tyler, Ph.D., University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01DC005972 (NIH); R01DC005972 (NIH)
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Other): Counseling plus everyday noise type 1
  Interventions: Other: Counseling and Sound Therapy
- 2 (Other): Counseling plus static noise type 2
  Interventions: Other: Counseling and Sound Therapy
- 3 (Other): Counseling plus static noise type 3
  Interventions: Other: Counseling and Sound Therapy
- 4 (Other): Hearing aid and counseling plus everyday noise type 1
  Interventions: Other: Counseling and Sound Therapy
- 5 (Other): Hearing aid and counseling plus static noise type 2
  Interventions: Other: Counseling and Sound Therapy
- 6 (Other): Hearing aid and counseling plus static noise type 3
  Interventions: Other: Counseling and Sound Therapy

INTERVENTIONS:
Other: Counseling and Sound Therapy — Tinnitus counseling and sound therapy

SUMMARY:
Millions of Americans suffer from tinnitus. However, there is no widely accepted treatment that has been shown to be effective in controlled investigations. The purpose of this study is to evaluate the effectiveness of Tinnitus Retraining Therapy (TRT). This study will investigate the contributions of counseling, the use of hearing aids and sound generators, and the importance of setting masking noise to a particular level. All groups will receive the same Counseling. In pilot studies we have developed a picture-based counseling protocol. The results of this study will determine if TRT is more effective than masking or counseling alone.

ELIGIBILITY:
Inclusion Criteria:

* Have experienced tinnitus for at least 4 months.
* Have the ability to participate in research.

Exclusion Criteria:

* Have a treatable otological disorder.
* Are involved in litigation.
* Have or are suspected of having a serious psychiatric problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2004-01; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Iowa Tinnitus Handicap Questionnaire | 18 months

SECONDARY OUTCOMES:
Tinnitus measures | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Tyler, Ph.D., Principal Investigator — University of Iowa
Locations (4):
- United States (4):
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - University at Buffalo, State University of New York, Buffalo, New York
  - East Tennessee State University, Johnson City, Tennessee